CLINICAL TRIAL: NCT03414658
Title: A Randomized, Phase II Study Comparing Trastuzumab and Vinorelbine in Combination With Avelumab or Avelumab and Utomilumab (41BB/CD137 Agonist), in Patients With HER2-positive Metastatic Breast Cancer Who Have Progressed on Prior Trastuzumab and Pertuzumab
Brief Title: The AVIATOR Study: Trastuzumab and Vinorelbine With Avelumab OR Avelumab & Utomilumab in Advanced HER2+ Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adrienne G. Waks (Other)
Collaborators: Pfizer (Industry); Breast Cancer Research Foundation (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Adrienne G. Waks, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-455; TBCRC045 (Other: TBCRC)
Record Dates: First submitted 2017-11-10; First posted 2018-01-30 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Trastuzumab; avelumab; utomilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NH: Trastuzumab + Vinorelbine (Experimental): * Trastuzumab is administered intravenously twice per cycle
  * Vinorelbine is administered intravenously 3 times per cycle
  Interventions: Drug: Vinorelbine; Drug: Trastuzumab
- NHA: Trastuzumab + Vinorelbine + Avelumab (Experimental): * Trastuzumab is administered intravenously twice per cycle
  * Vinorelbine is administered intravenously 3 times per cycle
  * Avelumab is administered intravenously twice per cycle
  * Antihistamine and with acetaminophen is mandatory 30 to 60 minutes prior to each dose of avelumab
  Interventions: Drug: Vinorelbine; Drug: Trastuzumab; Drug: Avelumab
- NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab (Experimental): * Trastuzumab is administered intravenously twice per cycle
  * Vinorelbine is administered intravenously 3 times per cycle
  * Avelumab is administered intravenously twice per cycle
  * Antihistamine and with acetaminophen is mandatory 30 to 60 minutes prior to each dose of avelumab
  * Utomilumab is administered intravenously once per cycle
  Interventions: Drug: Vinorelbine; Drug: Trastuzumab; Drug: Avelumab; Drug: Utomilumab

INTERVENTIONS:
Drug: Vinorelbine — work by interfering with cell division, which leaves the tumor unable to grow and spread
Drug: Trastuzumab — trastuzumab induces an antibody-dependent cell-mediated cytotoxicity against tumor cells that overexpress HER2.
Drug: Avelumab — monoclonal antibody directed against the human immunosuppressive ligand programmed death-ligand 1 (PD-L1) protein
  Arms: NHA: Trastuzumab + Vinorelbine + Avelumab; NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab
Drug: Utomilumab — Utomilumab is an antibody designed to stimulate the body's immune system to fight cancer cells
  Arms: NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for breast cancer.

The drugs involved in this study are:

* Group A: Trastuzumab (Herceptin) + Vinorelbine (Navelbine)
* Group B: Trastuzumab + Vinorelbine + Avelumab
* Group C: Trastuzumab + Vinorelbine + Avelumab + Utomilumab (PF-05082566)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug combination to learn whether the drug combination works in treating a specific disease. "Investigational" means that drug combination is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Utomilumab as a treatment for any disease.

The FDA (the U.S. Food and Drug Administration) has approved Avelumab as a treatment for other diseases.

The FDA (the U.S. Food and Drug Administration) has approved trastuzumab as a treatment option for this disease.

The FDA (the U.S. Food and Drug Administration) has approved vinorelbine as a treatment for other diseases and is commonly used as a treatment option for this disease.

The immune system is the body's natural defense against disease. The immune system sends a type of cells called T cells throughout the body to detect and fight infections and diseases-including cancers. One way the immune system controls the activity of T cells is through the PD-1 (programmed cell death protein-1) pathway. However, some cancer cells hide from T-cell attack by taking control of the PD-1 pathway and this stops T cells from attacking cancer cells. Avelumab is a type of drug, known as an antibody which is designed to block the PD-1 pathway and helps the immune system in detecting and fighting cancer cells. An antibody is a protein produced by the body's immune system when it detects harmful substances. Previous studies show that the administration of antibodies which block the PD-1 pathway can lead to tumor destruction.

Utomilumab is an antibody designed to stimulate the body's immune system to fight cancer cells. Previous studies have shown that the administration of this type of antibody may help to prevent tumors from growing.

In the laboratory, adding avelumab and Utomilumab to trastuzumab appears to improve effectiveness. It is not known whether this is true in humans.

In this research study, the investigators are evaluating the activity of 3 different combinations: (a)trastuzumab and vinorelbine combined, (b) trastuzumab, vinorelbine and avelumab combined, and (c) trastuzumab, vinorelbine, avelumab and utomilumab combined in participants with metastatic HER2- positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or older
* Histologically confirmed breast adenocarcinoma that is unresectable loco-regionally advanced or metastatic
* HER2-positive (immunohistochemistry score 3+) or ERBB2- amplification (Ratio ERBB2/centromeres ≥ 2.0 or mean gene copy number ≥ 6) on primary tumor or of metastatic or unresectable loco-regional biopsy.
* Measurable disease per RECIST v1.1 (see Section 11)
* Patients must have previous treatment with ado-trastuzumab emtansine (Kadcyla, T-DM1) in any setting. Patients must have previously received trastuzumab and pertuzumab in the metastatic setting or within 12 months of neoadjuvant/adjuvant treatment.
* Patient must have progressed on their most recent line of therapy. Progression must have been demonstrated by radiological or clinical assessment.
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Willingness and availability to submit FFPE tissue for central confirmation of HER2 positivity and central assessment of PD-L1 status. This can be from archival tissue from unresectable loco-regional or metastatic disease obtained ≤ 1 year prior to enrollment or new tissue material from a recently obtained surgical or diagnostic biopsy. Tissue obtained for the biopsy must not have been previously irradiated. If a patient does not have any available archival tissue ≤ 1 year old and the treating investigator does not feel that it would be safe to perform a fresh biopsy, the requirement for a fresh biopsy may be waived after discussion with the Principal Investigator.
* Written informed consent for screening and trial participation procedures including biological material transfer and handling.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Hematopoietic status:

  * Absolute neutrophil count ≥ 1.0 × 109/L,
  * Platelet count ≥ 100 × 109/L,
  * Hemoglobin ≥ 9 g/dL
* Hepatic status:

  * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN). In the case of known Gilbert's syndrome, a higher serum total bilirubin (< 2 × ULN) is allowed.
  * AST and ALT ≤ 2.5 × ULN; if the patient has liver metastases, ALT and AST must be ≤ 5 × ULN.
* Renal status:

  * Creatinine ≤ 1.5 ×ULN or creatinine clearance > 60 ml/min
  * Proteinuria < 1 g/day
* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulant.
* If female of childbearing potential, must have a negative pregnancy test within 7 days of initiating treatment. Childbearing potential is defined by: those who have not been surgically sterilized and/or have had a menstrual period in the past year.
* Participants of childbearing potential (as defined above) must be willing to use effective contraception during treatment and up to 7 months after stop of trial treatment. Acceptable methods of contraception are intrauterine devices, bilateral tubal occlusion, vasectomized, or total abstinence. Oral, injectable, or implant hormonal contraceptives are not allowed.
* Must not be breastfeeding/lactating.

Exclusion Criteria:

* Prior therapy with any anti-PD-1, anti-PD-L1, L2, anti-4-1BB (CD137), or anti-CTLA4 therapy
* Known Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Positive for Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA [qualitative]).
* History of interstitial lung disease
* Active central nervous system metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (patients with history of CNS metastases or spinal cord compression are eligible if they are clinically stable for at least 4 weeks before first dose of investigational product and do not require high-dose steroid treatment).
* History of clinically significant or uncontrolled cardiac disease, including congestive heart failure (New York Heart Association functional classification ≥3), angina, myocardial infarction or ventricular arrhythmia.
* Previous severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Active infection requiring systemic therapy.
* Chronic systemic therapy with immunosuppressive agents including corticosteroids.
* Active autoimmune disease or a documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the trial. Patients with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the trial.
* Concurrent disease or condition that would make the patient inappropriate for trial participation or any serious medical disorder that would interfere with the patient's safety.
* No uncontrolled hypertension (≥180/110), unstable diabetes mellitus, dyspnea at rest, or chronic therapy with oxygen.
* Chemotherapy, radiotherapy, and/or biological cancer therapy within 3 weeks prior to the first trial dose or has not recovered to CTCAE v.4 grade 1 or better from adverse events (except alopecia).
* Unresolved or unstable, serious adverse events from prior administration of another investigational drug.
* Live vaccines within 30 days prior to the first dose of trial therapy and during trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2026-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Waks, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Fred Hutchinson Cancer Care, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: AVIATOR enrolled 100 patients in 16 centers in the US between June 21, 2018 and March 1, 2023.
Groups:
- NH: Trastuzumab + Vinorelbine: * Trastuzumab is administered intravenously twice per cycle
  * Vinorelbine is administered intravenously 3 times per cycle
  Vinorelbine: work by interfering with cell division, which leaves the tumor unable to grow and spread
  Trastuzumab: trastuzumab induces an antibody-dependent cell-mediated cytotoxicity against tumor cells that overexpress HER2.
- NHA: Trastuzumab + Vinorelbine + Avelumab: * Trastuzumab is administered intravenously twice per cycle
  * Vinorelbine is administered intravenously 3 times per cycle
  * Avelumab is administered intravenously twice per cycle
  * Antihistamine and with acetaminophen is mandatory 30 to 60 minutes prior to each dose of avelumab
  Vinorelbine: work by interfering with cell division, which leaves the tumor unable to grow and spread
  Trastuzumab: trastuzumab induces an antibody-dependent cell-mediated cytotoxicity against tumor cells that overexpress HER2.
  Avelumab: monoclonal antibody directed against the human immunosuppressive ligand programmed death-ligand 1 (PD-L1) protein
- NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab: * Trastuzumab is administered intravenously twice per cycle
  * Vinorelbine is administered intravenously 3 times per cycle
  * Avelumab is administered intravenously twice per cycle
  * Antihistamine and with acetaminophen is mandatory 30 to 60 minutes prior to each dose of avelumab
  * Utomilumab is administered intravenously once per cycle
  Vinorelbine: work by interfering with cell division, which leaves the tumor unable to grow and spread
  Trastuzumab: trastuzumab induces an antibody-dependent cell-mediated cytotoxicity against tumor cells that overexpress HER2.
  Avelumab: monoclonal antibody directed against the human immunosuppressive ligand programmed death-ligand 1 (PD-L1) protein
  Utomilumab: Utomilumab is an antibody designed to stimulate the body's immune system to fight cancer cells
Period: Overall Study
Arm/Group | NH: Trastuzumab + Vinorelbine | NHA: Trastuzumab + Vinorelbine + Avelumab | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab
Started | 20 | 46 | 34
Completed | 18 | 45 | 34
Not Completed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NH: Trastuzumab + Vinorelbine | NHA: Trastuzumab + Vinorelbine + Avelumab | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab | Total
Number analyzed (Participants) | 18 | 45 | 34 | 97
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [44 to 60] | 53 [48 to 60] | 57 [46 to 63] | 54 [46 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 45 | 33 | 96
  Male | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 6 | 1 | 7
  Not Hispanic or Latino | 18 | 38 | 31 | 87
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 4 | 14
  White | 11 | 31 | 26 | 68
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 1 | 2 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 18 | 45 | 34 | 97
ECOG PS [Count of Participants; unit: Participants] — The ECOG Performance Status Scale is a measurement used to assess how cancer impacts a patient's daily living abilities. Smaller grades are considered better outcomes, eg. grade 0 means "fully active, able to carry on all pre-disease performance without restriction."
  Participants
    0 | 11 | 24 | 23 | 58
    1 | 7 | 21 | 11 | 39
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 23.8 [20.9 to 29.7] | 24.9 [23.1 to 27.8] | 26.4 [23.7 to 29.3] | 25.2 [22.5 to 29.1]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free Survival is defined from the time from randomization to the first occurrence of disease progression as determined by the investigator using RECIST 1.1 or death from any cause, whichever occurs first.
Time Frame: 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | NH: Trastuzumab + Vinorelbine | NHA: Trastuzumab + Vinorelbine + Avelumab | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab
Number analyzed (Participants) | 18 | 45 | 34
months | 2 [1.7 to 3.9] | 3.8 [3 to 5.5] | 4.9 [3.7 to 5.5]
Statistical Analysis 1: Comparison: NH: Trastuzumab + Vinorelbine vs NHA: Trastuzumab + Vinorelbine + Avelumab; Test type: Superiority; p = 0.025, Log Rank; Hazard Ratio (HR) = 0.53, 80% CI 2-sided [0.35 to 0.81]
Statistical Analysis 2: Comparison: NHA: Trastuzumab + Vinorelbine + Avelumab vs NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab; Test type: Superiority; p = 0.32, Log Rank; Hazard Ratio (HR) = 1.14, 80% CI 2-sided [0.8 to 1.64]

2. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate is determined by Complete Response or Partial Response by RECIST 1.1. Per RECIST 1.1 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Number (90% Confidence Interval); unit: percent of participants
Arm/Group | NH: Trastuzumab + Vinorelbine | NHA: Trastuzumab + Vinorelbine + Avelumab | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab
Number analyzed (Participants) | 18 | 45 | 34
percent of participants | 11.1 [2 to 31] | 20 [10.9 to 32.3] | 11.8 [4.1 to 24.9]

3. Secondary Outcome: Duration of Response
Description: Duration of Response is measured from the time criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Per RECIST 1.1 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 3 years
Population: Participants who had response.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | NH: Trastuzumab + Vinorelbine | NHA: Trastuzumab + Vinorelbine + Avelumab | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab
Number analyzed (Participants) | 2 | 9 | 4
months | NA [NA to NA] — Values are NA due to insufficient number of participants with events: only 2 patients had response in NH arm. The DOR of them are 4 and 10.3 months. | 15.8 [3.6 to 25.2] | 4.2 [3 to NA] — 90% UCL could not be estimated due to insufficient number of participants with event.

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death from any cause, or is censored at date last known alive.
Time Frame: 5 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | NH: Trastuzumab + Vinorelbine | NHA: Trastuzumab + Vinorelbine + Avelumab | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab
Number analyzed (Participants) | 18 | 45 | 34
months | 22.8 [17.4 to NA] — 90% UCL could not be estimated due to insufficient number of participants with events. | 26.3 [15.9 to 36.1] | 27 [17.3 to 33.7]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality measurement is assessed every 8-12 weeks during treatment. After protocol therapy then assessed annually until death, withdrawal of consent, or lost to follow-up. The observed maximum follow up 52 months (from overall survival). Adverse events(SAEs and OAEs) are assessed every 8-12 weeks. After protocol therapy, assessed approximately 4 weeks following completion of therapy. The median(range) number of competed cycles of therapy was 4(1-34). As such up to 136 weeks.
Description: A serious adverse event (SAE) is an undesirable sign, symptom, or medical condition which:is fatal;is life-threatening;requires or prolongs inpatient hospitalization for ≥24 hours;results in persistent or significant disability/incapacity to conduct normal life functions;constitutes a congenital anomaly or birth defect; or jeopardizes the participant and requires medical or surgical intervention to prevent one of the outcomes listed above; Remaining AEs are classified as Other AEs (OAEs).
Arm/Group | NH: Trastuzumab + Vinorelbine | NHA: Trastuzumab + Vinorelbine + Avelumab | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab
All-Cause Mortality (participants affected / at risk) | 10/18 | 23/45 | 20/34
Serious Adverse Events (participants affected / at risk) | 5/18 | 9/45 | 9/34
Other Adverse Events (participants affected / at risk) | 18/18 | 45/45 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NH: Trastuzumab + Vinorelbine (N=18) | NHA: Trastuzumab + Vinorelbine + Avelumab (N=45) | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab (N=34)
Death NOS (General disorders) | 1 | 0 | 0
Fever (General disorders) | 2 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Lung infection (Infections and infestations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Serum amylase increased (Investigations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NH: Trastuzumab + Vinorelbine (N=18) | NHA: Trastuzumab + Vinorelbine + Avelumab (N=45) | NHAU: Trastuzumab + Vinorelbine + Avelumab + Utomilumab (N=34)
Anemia (Blood and lymphatic system disorders) | 11 | 17 | 15
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 3 | 11 | 4
Blurred vision (Eye disorders) | 1 | 3 | 2
Cataract (Eye disorders) | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 1
Dry eye (Eye disorders) | 1 | 4 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 3 | 1
Eye pain (Eye disorders) | 1 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 1 | 0
Floaters (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Watering eyes (Eye disorders) | 0 | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 7 | 10
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 3 | 3 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Colonic ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 8 | 17 | 16
Diarrhea (Gastrointestinal disorders) | 4 | 10 | 10
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 5 | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 6 | 5
Nausea (Gastrointestinal disorders) | 9 | 17 | 15
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 2 | 8
Chills (Gastrointestinal disorders) | 0 | 4 | 0
Edema face (General disorders) | 0 | 1 | 1
Edema limbs (General disorders) | 4 | 0 | 2
Fatigue (General disorders) | 15 | 28 | 27
Fever (General disorders) | 3 | 3 | 3
Flu like symptoms (General disorders) | 1 | 3 | 2
Gait disturbance (General disorders) | 1 | 2 | 0
General disorders and administration site conditions - Other, specify (Gastrointestinal disorders) | 1 | 4 | 3
Infusion related reaction (General disorders) | 1 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 0 | 1 | 0
Neck edema (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 2
Pain (General disorders) | 1 | 7 | 7
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 1
Autoimmune disorder (Immune system disorders) | 0 | 1 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 2 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1
Rhinitis infective (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 2
Skin infection (Infections and infestations) | 3 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 4 | 1
Urinary tract infection (Infections and infestations) | 1 | 6 | 2
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 2 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 10 | 4
Alkaline phosphatase increased (Investigations) | 2 | 11 | 5
Aspartate aminotransferase increased (Investigations) | 4 | 14 | 8
Blood bilirubin increased (Investigations) | 0 | 1 | 2
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1
Cholesterol high (Investigations) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 2 | 3
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Investigations - Other, specify (Investigations) | 0 | 2 | 3
Lipase increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 4 | 6
Neutrophil count decreased (Investigations) | 12 | 29 | 22
Platelet count decreased (Investigations) | 2 | 7 | 6
Serum amylase increased (Investigations) | 0 | 1 | 0
Weight gain (Investigations) | 1 | 2 | 0
Weight loss (Investigations) | 0 | 3 | 3
White blood cell decreased (Investigations) | 4 | 12 | 10
Anorexia (Metabolism and nutrition disorders) | 5 | 5 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 5 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 4
Hypokalemia (Metabolism and nutrition disorders) | 0 | 3 | 6
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 11 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 5 | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 4 | 4
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 5
Headache (Nervous system disorders) | 2 | 13 | 7
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 4 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 20 | 15
Presyncope (Nervous system disorders) | 0 | 1 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 3 | 4 | 11
Confusion (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 4 | 6
Insomnia (Psychiatric disorders) | 0 | 5 | 9
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 2 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 4 | 4 | 4
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Nipple deformity (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 2 | 2
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 2 | 1
Uterine obstruction (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 9 | 7
Body odor (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5 | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 6 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 2 | 4 | 4
Hot flashes (Vascular disorders) | 0 | 3 | 5
Hypertension (Vascular disorders) | 3 | 4 | 6
Hypotension (Vascular disorders) | 0 | 3 | 1
Lymphedema (Vascular disorders) | 1 | 5 | 3
Thromboembolic event (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT03414658/Prot_SAP_000.pdf